CLINICAL TRIAL: NCT03951038
Title: Efficacy and Safety of Ultrasound-guided Lateral Thoracolumbar Interfascial Plane Block (TLIPB) for Postoperative Pain in Patients Undergoing Herniated Lumbar Disc Surgery: A Randomized Clinical Trial.
Brief Title: Efficacy and Safety of Ultrasound-guided Lateral Thoracolumbar Interfascial Plane Block (TLIPB) for Postoperative Pain in Patients Undergoing Herniated Lumbar Disc Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Min Su, Clinical Professor, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CQMUAZD2019
Record Dates: First submitted 2019-05-08; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Postoperative Pain; Lumbar Disc Surgery
Keywords: Lumbar disc herniation; Postoperative analgesia; Patient controlled intravenous analgesia; Nerve block; thoracolumbar
MeSH Terms: conditions — Pain, Postoperative; Intervertebral Disc Displacement | interventions — Nerve Block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCIA group (Active Comparator): Participants in this group will receive PCIA post-operatively (tramadol 800 mg and flurbiprofen axetil 100mg with saline added up to a volume of 80ml in total ) and the equal volume of 0.9% normal saline will be conducted by ultrasound and receive a single injection between the longissimus and iliocostalis muscles both sides of the spine. The PCIA pump was set up with a 5 ml loading dose, a 2 ml bolus dose, a 15 min lockout interval and background infusion at a rate of 1 ml/h.
  Interventions: Procedure: PCIA group
- Lateral TLIPB group (Experimental): Participants in this group will be conducted by ultrasound and receive a single injection between the longissimus and iliocostalis muscles both sides of the spine, and combined with PCIA post-operatively. The regimen of the Lateral TLIPB is 0.2% 20 ml ropivacaine respectively and the regimen of PCIA is same with PCIA group.
  Interventions: Procedure: Lateral TLIPB group

INTERVENTIONS:
Procedure: PCIA group — The formula of the PCIA included tramadol 800 mg, flurbiprofen axetil 100mg with saline added up to a volume of 80 ml in total. The PCIA pump was set up with a 5 ml loading dose, a 2 ml bolus dose, a 15 min lockout interval and background infusion at a rate of 1 ml/h.
  Arms: PCIA group
Procedure: Lateral TLIPB group — both sides of the spine, a single injection of ropivacaine by nerve stimulating needle under ultrasound-guided between the longissimus and iliocostalis muscles .
  The regimen of Lateral TLIPB group is0.2% 20ml ropivacaine and the regimen of PCIA is same with PCIA group.
  Other Names: Nerve block
  Arms: Lateral TLIPB group

SUMMARY:
Surgery of the lumbar spine is characterized by diffuse and severe postoperative pain. In recent years, some case reports indicate that the thoracolumbar interfascial plane block (TLIPB) can reduce postoperative pain after spinal surgery, which targets the dorsal roots of the thoracolumbar nerves by depositing local anesthetic at the level of third lumbar vertebra between the multiﬁdus and longissimus muscles. However, a new approach of the TLIPB technique by injecting local anesthetic between the longissimus and iliocostalis muscles, that is the Lateral TLIPB. According some relevant literature reports show that this technique simpler to perform and reduces the risk of neuraxial puncture. So, the purpose of this study is to investigate the efficacy and safety of the Lateral TLIPB combined with patient controlled intravenous analgesia (PCIA) is superior to PCIA in reducing postoperative pain in patients undergoing spinal surgery.

DETAILED DESCRIPTION:
Although the number of spinal surgeries has been increasing for many years, the methods for perioperative pain relief have remained limited. According to some report show that surgery of the lumbar spine is characterized by diffuse and severe postoperative pain. Pre/postoperative oral opioids, gabapentinoids, nonsteroidal antiinﬂammatory drugs are frequently included in multimodal analgesia for spinal surgery, but the effect was not satisfactory. The ultrasound-guided thoracolumbar interfascial plane block (TLIPB) is a peripheral nerve block, which injecting local anesthetic between the muitifidus and longissimus muscles at the level of 3rd lumbar vertebra and can block the dorsal rami of thoracolumbar nerves. TLIPB have the potential to provide long-lasting postoperative analgesia and reduce opioid consumption while minimizing the motor block associated with neuraxial and plexus blocks. However, a new approach of the TLIPB technique by injecting local anesthetic between the longissimus and iliocostalis muscles, that is the Lateral TLIPB. Comparing with the TLIPB, Lateral TLIPB have some advantages, first; ultrasonographic identiﬁcation of the multiﬁdus and longissimus muscles may be difﬁcult, and it is easier to find the plane between the longissimus and iliocostal muscles, so, the success rate of puncture is higher; secondly; lateral to medial needle advancement can cause inadvertent neuroaxial puncture. A medial to lateral approach may be safer to perform to avoid dural puncture. So, the purpose of this study is to investigate the efficacy and safety of the Lateral TLIPB combined with patient controlled intravenous analgesia (PCIA) is superior to PCIA in reducing postoperative pain in patients undergoing spinal surgery.

This study was approved by the institutional review board of the First Affiliated Hospital of Chongqing Medical University. The protocol design is in accordance with Consolidated Standards of Reporting Trials (CONSORT) statement. All potentially eligible participants will be asked to give written informed consent before they are enrolled in this study. This study is a prospective, randomized, double-blind, controlled clinical trial guided by the standard of good clinical practice (GCP), and eligible participants are divided into two groups: group Lateral TLIPB and group PCIA, and primary assess the outcomes of the intensity of acute pain after Lumbar disc surgery.

Participants in group Lateral TLIPB will receive a single injection local anesthetic at the level of third lumbar vertebra between the longissimus and iliocostalis muscles on either side of the spine, and combined with PCIA post-operatively.

Participants in group PCIA will receive the equal volume of 0.9% normal saline between the longissimus and iliocostalis muscles on either side of the spine and PCIA post-operatively.

The primary outcome of this study is the intensity of acute pain after Lumbar disc surgery.The secondary outcomes of this study rescue medication and adverse events associated with the post-operative analgesia.

This study will be conducted under the supervision of an independent auditor. Every week, the auditor checked the data of the participants the day after the surgery was conducted. Assessment of pain intensity and prognostic outcomes must be confirmed by the auditor in sample population. When there is disagreement between surgeon and anesthesiologists in evaluating the prognosis of patients, the auditor must solve this disagreement by discussion with evaluators. Data will be double-entered by two statisticians with limitation of access and locked during statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. men or woman and 18～65 years old
2. clinical diagnosis of umbar disc herniation and will receive selective Lumbar disc surgery

Exclusion Criteria:

1. age below 18 years or over 65 years;
2. American Society of Anesthesiologists grade III or greater;
3. Diabetes;
4. allergic to local anesthetics;
5. cognitive impairment or communication problems;
6. received opioids、NSAID or tranquilizers (treatment for over 1 wk before the surgery);
7. history of alcohol or drug abuse;
8. severe hepatic or renal impairment ;
9. post-operative severe complications(e.g. pyogenic infection)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-02-14 (Estimated)

PRIMARY OUTCOMES:
Acute pain post-operatively | 6 hours post-operatively
  Pain intensity will be measured by visual analogue scale(VAS)， which included an 11-point scale with 0 labeled as "no pain" and 10 as "worst possible pain". Pain intensity was classified as mild with scores of 1～3, moderate with scores of 4～6, and severe with scores of 7～10.
Acute pain post-operatively | 12 hours post-operatively
  Pain intensity will be measured by visual analogue scale(VAS)
Acute pain post-operatively | 24 hours post-operatively
  Pain intensity will be measured by visual analogue scale(VAS)
Acute pain post-operatively | 36 hours post-operatively
  Pain intensity will be measured by visual analogue scale(VAS)
Acute pain post-operatively | 48 hours post-operatively
  Pain intensity will be measured by visual analogue scale(VAS)

SECONDARY OUTCOMES:
Analgesic Rescue | post-operative day 1 to 2
  The dosages of opioid or non-opioid analgesic rescue medications
The number of pushed and requested PCA | post-operative day 1 to 2
Incidence of adverse events associated with post-operative analgesia | post-operative day 1 to 2
  Including inadequate analgesia; nausea and vomiting; respiratory depression; local infection

CONTACTS AND LOCATIONS:
Overall Officials: Su Min, MD, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Ahiskalioglu A, Yayik AM, Alici HA. Ultrasound-guided lateral thoracolumbar interfascial plane (TLIP) block: Description of new modified technique. J Clin Anesth. 2017 Aug;40:62. doi: 10.1016/j.jclinane.2017.04.015. No abstract available. PMID 28625449
- [Background] Ueshima H, Hara E, Otake H. RETRACTED: Thoracolumbar interfascial plane block provides effective perioperative pain relief for patients undergoing lumbar spinal surgery; a prospective, randomized and double blinded trial. J Clin Anesth. 2019 Dec;58:12-17. doi: 10.1016/j.jclinane.2019.04.026. Epub 2019 Apr 25. PMID 31029989 (Retraction: PMID 35393187 J Clin Anesth. 2022 Aug;79:110690)
- [Background] Li C, Jia J, Qin Z, Tang Z. The use of ultrasound-guided modified thoracolumbar interfascial plane (TLIP) block for multi-level lumbar spinal surgery. J Clin Anesth. 2018 May;46:49-51. doi: 10.1016/j.jclinane.2018.01.018. Epub 2018 Mar 26. No abstract available. PMID 29414616
- [Background] Ammar MA, Taeimah M. Evaluation of thoracolumbar interfascial plane block for postoperative analgesia after herniated lumbar disc surgery: A randomized clinical trial. Saudi J Anaesth. 2018 Oct-Dec;12(4):559-564. doi: 10.4103/sja.SJA_177_18. PMID 30429737
- [Background] Ahiskalioglu A, Yayik AM, Doymus O, Selvitopi K, Ahiskalioglu EO, Calikoglu C, Alici HA, Karaca O. Efficacy of ultrasound-guided modified thoracolumbar interfascial plane block for postoperative analgesia after spinal surgery: a randomized-controlled trial. Can J Anaesth. 2018 May;65(5):603-604. doi: 10.1007/s12630-018-1051-0. Epub 2018 Jan 9. No abstract available. PMID 29318534
- [Background] Manchikanti L, Helm Ii S, Singh V, Hirsch JA. Accountable interventional pain management: a collaboration among practitioners, patients, payers, and government. Pain Physician. 2013 Nov-Dec;16(6):E635-70. PMID 24284849
- [Background] Rajaee SS, Bae HW, Kanim LE, Delamarter RB. Spinal fusion in the United States: analysis of trends from 1998 to 2008. Spine (Phila Pa 1976). 2012 Jan 1;37(1):67-76. doi: 10.1097/BRS.0b013e31820cccfb. PMID 21311399
- [Background] Hand WR, Taylor JM, Harvey NR, Epperson TI, Gunselman RJ, Bolin ED, Whiteley J. Thoracolumbar interfascial plane (TLIP) block: a pilot study in volunteers. Can J Anaesth. 2015 Nov;62(11):1196-200. doi: 10.1007/s12630-015-0431-y. Epub 2015 Jul 7. PMID 26149600
- [Background] Ueshima H, Sakai R, Otake H. Clinical experiences of ultrasound-guided thoracolumbar interfascial plane block: a clinical experience. J Clin Anesth. 2016 Sep;33:499. doi: 10.1016/j.jclinane.2015.09.005. Epub 2015 Oct 23. No abstract available. PMID 26507177